CLINICAL TRIAL: NCT00889694
Title: Clinical Study of Tripterygium Capsule to Treat Early Ankylosing Spondylitis: a 12-Week, Multiple Centers, Randomized Double-Blind, Positive Drug and Placebo Controlled Clinical Trial
Brief Title: Clinical Study of Tripterygium Capsule to Treat Early Ankylosing Spondylitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Jieruo Gu, Rheumatology Department of Third Affiliated Hospital of Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: [2008]2-4
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Early Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Sulfasalazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tripterygium — Tripterygium: 2 capsules per time, 3 times per day for 12 weeks.
Drug: Sulfasalazine — Sulfasalazine: 0.75 gram per time, 2 times per day for 12 weeks.
Drug: placebo — Placebo: 2 capsules per time, 3 times per day for 12 weeks.

SUMMARY:
This study is a 12-week, randomized, placebo and positive drug controlled clinical trial to investigate whether tripterygium capsule is effective and safe in treating patients with ankylosing spondylitis. The investigators expect that the tripterygium capsule is more effective than placebo and has few adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfill the ESSG criteria for SpA and not fulfill any criteria for the subtype including ankylosing spondylitis, psoriatic arthritis, reactive arthritis and inflammatory bowel disease associated arthritis.
2. Disease is in active status defined by BASDAI>=40mm.
3. DMARDs administration must be suspended for at least 4 weeks before screening. NSAIDs dose must be stable for at least 4 weeks before screening.

Exclusion Criteria:

1. Intra-articular injection of glucocorticoid within 3 months.
2. Previous history of heart failure, multiple sclerosis, chronic obstructive pulmonary disease, recurrent infection, lymphoma or other tumors.
3. Accompanied by fibromyalgia syndrome or other rheumatic diseases.
4. Female of pregnancy or breast-feeding.
5. Poor compliance or with mental diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-07 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
ASAS20 | 12th week

SECONDARY OUTCOMES:
BASDAI20/50/70 | 12th week